CLINICAL TRIAL: NCT03122964
Title: Multi Institutional Study To Evaluate Dna Methlyation Markers For Detection Of Primary Bladder Cancer In Urine Samples From A Cohort Of Patients With Hematuria
Brief Title: Multi Institutional Study in Patient Presenting With Hematuria
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: MDx Health (Industry)
Responsible Party: Sponsor
Other Study IDs: Hematuria
Record Dates: First submitted 2017-04-12; First posted 2017-04-21 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Bladder Cancer; Hematuria
MeSH Terms: conditions — Urinary Bladder Neoplasms; Hematuria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with gross or microscopic hematuria: This study aims to prospectively enroll a minimum of 700 subjects, with gross or microscopic hematuria. Each site will target enrollment of 100 subjects and patient samples will be collected from consecutive patients meeting the inclusion criteria outlined below. The total study duration is expected to be 24 months.
  Interventions: Diagnostic Test: AssureMDx

INTERVENTIONS:
Diagnostic Test: AssureMDx — combined panel of methylation and mutation markers for the detection of bladder cancer

SUMMARY:
The primary objective of this study is to evaluate the performance of the methylation marker panel for the detection of bladder cancer in patients with gross or microscopic hematuria.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the performance of the methylation marker panel for the detection of bladder cancer in patients with gross or microscopic hematuria.

The secondary objective is to evaluate the predictive accuracy of a risk model including clinical factors such as age, gender, smoking history, and presence of gross versus microscopic hematuria compared to a model incorporating the same risk factors along with the methylation marker panel.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is willing and able to give written informed consent
2. Subject presents with or has a history of gross hematuria or microhematuria within the last 3 months

Exclusion Criteria:

1. Subject has an active urinary tract infection, current urinary retention, active stone disease (renal or bladder), current ureteral stents or nephrostomy tubes, prior bowel interposition, or recent genitourinary instrumentation (within 10 days)
2. Subject has a current or past history of genitourinary or urologic cancer within 5 years
3. Subject has an active (untreated) cancer of any type, except basal cell skin cancer within 5 years

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subject presents with or has a history of gross hematuria or micro hematuria within the last 3 months
Sampling Method: Non-Probability Sample
Enrollment: 1148 (Actual)
Dates: Start 2017-03-31 (Actual); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Performance of a panel of methylation markers for the detection of bladder cancer in patient presenting with hematuria. | 1 year
  Early detection of bladder cancer in patients presenting with hematuria

SECONDARY OUTCOMES:
Predictiveness of a panel of methylation markers combined with clinical risk factors for the detection of bladder cancer. | 1 year
  Accurately predict clinical risk of bladder cancer through clinical factors and methylation markers

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No